CLINICAL TRIAL: NCT04331223
Title: The Association of Clinical Symptom Clusters With Underlying Mechanisms in Functional Gastrointestinal Disorders
Status: Completed | Type: Observational
Sponsor: Brain-Gut Research Group (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DK5
Record Dates: First submitted 2018-12-14; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Irritable Bowel Syndrome; Functional Dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — observational

SUMMARY:
Functional gastrointestinal disorders (FGID) are amongst the most common causes of abdominal pain and dysfunction seen in clinical practice, affecting between 10 to 15% of most populations (1). FGID are defined by symptoms without demonstrable underlying organic pathology (2). Within the currently used Rome definitions of FGID, there is a broad range of gastrointestinal and multi-organ symptoms, indicating heterogeneous underlying pathophysiological mechanisms (3). There is evidence of central nervous system and motility dysfunction, dysbiosis, as well as immune activation in various subgroups of patients with FGID (2). Most mechanistic studies have been performed in small and heavily selected groups of patients. Consequently, the link between different symptomatic subgroups of patients and underlying mechanisms is unclear and unconfirmed in larger and representative patient cohorts. FGID patients with different underlying pathologies are likely to benefit from divergent specific treatments, even if they fall within the same Rome classification of FGID.

Discrete clusters of clinical characteristics in a large cohort of patients with FGID will be sought using hypothesis-free cluster analysis and latent-class analysis models. Associations to underlying mechanisms will be examined using data from fermentable sugar breath, blood and stool tests. This will allow recommendations regarding improved mechanistic-based classifications of patients with FGID, with potential for more effective mechanistic-based treatments.

The investigators will use coded clinical and medical history characteristics obtained by standardized questionnaires and laboratory and breath test results from all successive patients above the age of 18 years referred to the Gastroenterology Group Practice in the last 10 years for diagnosis and treatment of FGID for statistical analysis The data is stored in a database, without any personal identifiers. Explorative statistical analysis will be performed in approximately 5000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Have FGID at time of referral based on Rome III criteria
* Age over 18 years

Exclusion Criteria:

* Evidence of organic disease.
* Age below 18 years
* Documented refusal to allow data use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male and female patients classified as having FGID at time of referral, based on Rome III criteria, and age over 18 years
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Clusters of clinical symptoms in Rome III Functional GI disorders assessed by Likert scale and defined by latent class analysis. | 6 months
  Clusters defined by latent class modelling of the most commonly reported symptoms assessed by Likert scale (3-point numerical rating scale ranging from 'none' to 'severe').

SECONDARY OUTCOMES:
Association of clusters (primary outcome) with demographic patient characteristics. | 6 months
  Association of clinical symptom cluster(primary outcome) with demographic patient characteristics.
Association of clusters (primary outcome) with gas concentrations during fructose and lactose breath test variables. | 6 months
  Testing of the association of clusters (primary outcome) with breath hydrogen, methane following fructose and lactose breath tests.
Association of clusters (primary outcome) with symptoms fructose and lactose breath test variables. | 6 months
  Testing of the association of clusters (primary outcome) with symptoms rated by Likert scale (3-point numerical rating scale ranging from 'none' to 'severe') following fructose and lactose breath tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastoenterology Group Practice; Brain-Gut Research Group, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No